CLINICAL TRIAL: NCT03042754
Title: Improve Treatment Outcomes for Tuberculosis Infection in Tertiary Care Hospitals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Bamrasnaradura Infectious Diseases Institute (Other Government); Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TB NRU
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis
Keywords: LAM; XpertMTB/RIF; treatment outcome; Microbacterial tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- suspected TB (Other): Patients suspected with TB will be sent for XpertMTB/RIF and urine LAM test
  Interventions: Diagnostic Test: XpertMTB/RIF

INTERVENTIONS:
Diagnostic Test: XpertMTB/RIF

SUMMARY:
Early diagnosis can contribute to good treatment outcomes and isolate infection control.

DETAILED DESCRIPTION:
This study is conducted into 2 parts: prospective and retrospective.

The prospective study evaluated the use of Xpert MTB/RIF. The study was conducted at three large tertiary care hospitals: the King Chulalongkorn Memorial Hospital, Rajavithi Hospital and Bamrasnaradura Infectious Diseases Institute. Only pulmonologists and infectious disease physicians with extensive experience in TB participated in the study. Patients who had suspected PTB were enrolled into the study. Expectorated sputum were collected and transferred to the central laboratory, Chulalongkorn Research Center (CRC) Laboratory, King Chulalongkorn Memorial Hospital. Each sample was divided into two parts; one part for the Xpert MTB/RIF (Cepheid) and another part for mycobacterial culture. Drug susceptibility tests for streptomycin, isoniazid, rifampicin and ethambutol were performed with rapid qualitative procedure (BACTEC™ MGIT™ 960 SIRE Kit) and semi-automated system (BACTEC™ MGIT™ 960 System). Discordant results of MGIT and Xpert were retested with the rpoB gene sequencing system. All PTB patients were promptly treated with anti-TB drug regimens as WHO's recommendation. All patients had HIV testing done and CD4 cell counts were obtained for all HIV-infected patients. Antiretroviral treatment and prophylaxis for opportunistic infections were prescribed as standard treatment guideline for patients with HIV/TB co-infection. The patients were followed until completion of TB treatment or change in the diagnosis. The WHO definitions for cure, completed treatment, dead, default or treatment failure were used to define the outcome of treatment.

The authors , therefore, evaluated the utility of Xpert MTB/RIF in Thailand, prior to nation-wide implementation. In summary, our real-life cohort study use Xpert MTB/RIF for early diagnosis of PTB and rifampicin resistance in high TB burden country outside of the African region. The results may be beneficial for guiding the policy makers, especially the National Tuberculosis Programme (NTP) to control TB transmission, as the country move towards universal use of Xpert MTB/RIF.

The retrospective study assessed the urine LAM test which has not been evaluated in non-HIV-infected immunocompromised Asians with disseminated TB and non-disseminated TB (TB located in one organ) but has a poor sensitivity and specificity for detecting pulmonary TB patients without HIV infection. On that account, the authors evaluated the applicability and efficacy of TB diagnosis by using the urine from confirmed cultured TB cases with various immune response conditions, such as HIV-infected, non-HIV-infected and non-HIV-infected immunocompromised patients. The authors found that the sensitivity of the urine LAM in HIV-infected and non-HIV-infected patients were similar to previous reports. This confirmed that the urine LAM cannot be used alone to screen for TB. However, it can be used in conjunction with the culture and AFB smear test for patients co-infected with HIV with very low CD4 count. The urine LAM test is especially helpful in cases where the smear is negative in probable-TB patients. For this reason, the urine LAM test is attractive because it is not invasive, and the samples needed can be easily collected from these types of disseminated patients with and without HIV.

Aside from that, the urine LAM test can be used in those severely ill patients, regardless of HIV infection, where it is difficult to physically collect the sputum and paucibacillary samples. The PPV was over 80% for those infected with HIV and up to 100% in non-HIV-infected patients. For physicians, the PPV is more useful than the sensitivity and specificity of the assay because it will answer the question how likely the patient with a positive result from the urine LAM test will have TB or not. A high PPV can accurately guide the physicians to confidentially prescribe the TB medications which are crucial, especially among co-infected patients that are severely ill. For this reason, the urine LAM test seems to be a great point-of-care test that can easily be incorporated with the AFB smear and culture test for the Asian population. Furthermore, this study demonstrated that a positive urine LAM test result was significantly associated with death, especially those with HIV infection. This association is much stronger in patients with very low CD4 counts. The findings from this study suggest the possible use of the urine LAM test with the AFB smear and culture in resource-limited countries in diagnosing TB in advanced HIV and non-HIV-infected patients with TB. This promising diagnostic tool can increase the yield of TB diagnosis and predict the mortality rate of TB infection, particularly in advanced HIV patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected TB
* patients that can give us sputum and urine specimens

Exclusion Criteria:

* refuse to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-06-06 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of sputum from patients suspected with TB | 2 years
Sensitivity of urine LAM from patients suspected with TB | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gompol Suwanpimolkul, MD, Principal Investigator — Chulalongkorn University; Kamon Kawkitinarong, MD, Principal Investigator — Chulalongkorn University
Locations (4):
- Thailand (4):
  - Chulalongkorn University, Bangkok
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - Rajavithi Hospital, Bangkok
  - Bamrasnaradura Institute, Nonthaburi

IPD SHARING:
Plan to Share IPD: No
only for auditing/monitoring process as needed

REFERENCES:
- See also: Related Info — http://www.hivnat.org